Official Title: Phase I/IIa Dose Escalation Safety and Efficacy Study of Human

Embryonic Stem Cell-Derived Retinal Pigment Epithelium Cells
Transplanted Subretinally in Patients With Advanced Dry-Form Age-

Related Macular Degeneration (Geographic Atrophy)

NCT Number: NCT02286089

**Document Date:** SAP version 1.0: 12-October-2022



## Statistical Analysis Plan (SAP) for

Phase I/IIa Dose Escalation Safety and Efficacy Study of Human Embryonic Stem Cell-Derived Retinal Pigment Epithelium Cells Transplanted Subretinally in Patients with Advanced Dry-Form Age-Related Macular Degeneration (Geographic Atrophy)

| Clinical Phase: | I/IIa |
|-----------------------------------|---------------------------------|
| Sponsor Details: | Lineage Cell Therapeutics, Inc. |
| | 2173 Salk Avenue, Suite 200 |
| | Carlsbad, CA 92008 USA |
| Protocol Number: | CCN_CT02 |
| Amendment number | 14 |
| Dated: | 9 April 2019 |
| Issue: | FINAL |
| www.ClinicalTrials.gov Identifier | NCT02286089 |
| SAP document version | 1.0 |
| Document date | 12 October 2022 |

#### **CONFIDENTIALITY STATEMENT**

The information in this document is considered the property of the Sponsor and is privileged and confidential. No unpublished information contained herein may be disclosed without prior written approval from the Sponsor. Access to this document must be restricted to relevant parties.

# Approval of Statistical Analysis Plan for Clinical Research Protocol No. CCN\_CT02 – Amendment #14

Phase I/IIa Dose Escalation Safety and Efficacy Study of Human Embryonic Stem Cell-Derived Retinal Pigment Epithelium Cells Transplanted Subretinally in Patients with Advanced Dry-Form Age-Related Macular Degeneration (Geographic Atrophy)

## Approved by:



Lineage Cell Therapeutics, Inc.
OpRegen® Protocol: CCN\_CT02 (Amendment #14)
Statistical Analysis Plan Version 1.0

12 October 2022

# **VERSION HISTORY**

| Version | Date | Status/Reason for Changes |
|---------|-----------------|---------------------------|
| 1.0 | 12 October 2022 | Initial Draft |

# **TABLE OF CONTENTS**

| 1.0 LIST OF ABBREVIATIONS | 6 |
|---|---|
| 2.0 INTRODUCTION | 8 |
| 3.0 STUDY OBJECTIVES AND ENDPOINTS | 8 |
| 3.1.1 Primary Objectives | 8 |
| 3.2 Study Endpoints | 9<br>9<br>9 |
| 3.3 Study Hypothesis | 10 |
| 3.4 Study Assessments Schedules | 10 |
| 4.0 STUDY DESIGN | 13 |
| 4.1 Definitions | 14 |
| 5.0 STUDY POPULATION | |
| 6.0 STATISTICAL ANALYSIS GENERAL CONSIDERATIONS | 15 |
| 6.1 Analysis Sets | 15 |
| 6.2 Significance Level | 16 |
| 6.3 Procedures for Handling Missing Data and Outliers | 16 |
| 6.4 Descriptive Statistics | 16 |
| 7.0 STATISTICAL METHODS | 16 |
| 7.1 Study Subjects 7.1.1 Subject Disposition. 7.1.2 Protocol Deviations. 7.1.3 Demographics. 7.1.4 Medical and Surgical History. 7.1.5 Concomitant Medications. 7.1.6 Adverse Events. 7.1.7 Clinical Laboratory Tests 7.1.8 Vital Signs. 7.1.9 Physical Exam. | |
| 7.1.10 Efficacy Analyses | |

| | ge Cell Therapeutics, Inc. | |
|--------|-------------------------------------------|-----------------|
| | egen® Protocol: CCN_CT02 (Amendment #14) | |
| Statis | tical Analysis Plan Version 1.0 | 12 October 2022 |
| 8.0 | GENERAL CONSIDERATIONS | |
| 9.0 | SEQUENCE OF PLANNED ANALYSES | 20 |
| 10.0 | REPORTING CONVENTIONS | 20 |
| 11.0 | SUMMARY TABLES, FIGURES AND DATA LISTINGS | 22 |

# 1.0 LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|---------------------------------------------|
| AE | Adverse Event |
| AMD | Age-Related Macular Degeneration |
| BCVA | Best Corrected Visual Acuity |
| CFP | Color Fundus Photography |
| CI | Confidence Interval |
| CNV | Choroidal Neovascularization |
| CRF | Case Report Form |
| CRP | C-Reactive Protein |
| CSR | Clinical Study Report |
| DLT | Dose-Limiting Toxicity |
| DSMB | Data Safety Monitoring Board |
| ESR | Erythrocyte Sedimentation Rate |
| EBV | Epstein-Barr Virus |
| ECG | Electrocardiogram |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| FA | Fluorescein Angiography |
| FAF | Fundus Autofluorescence (imaging) |
| FRI | Functional Reading Independence (FRI) Index |
| GA | Geographic Atrophy |
| GMP | Good Manufacturing Practice |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| hESCs | Human Embryonic Stem Cells |
| HLA | Human Leukocyte Antigen(s) |
| IB | Investigator's Brochure |
| IFU | Instructions for Use |
| IOP | Intraocular Pressure |
| LDH | Lactic Dehydrogenase |
| MedDRA | Medical Dictionary for Regulatory Affairs |
| MTD | Maximally Tolerated Dose |

12 October 2022

| Abbreviation | Definition |
|--------------|---------------------------------------------------------|
| NEI VFQ-25 | National Eye Institute Visual Function Questionnaire-25 |
| PP | Per Protocol |
| QoL | Quality of Life |
| RPE | Retinal Pigment Epithelium |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SD-OCT | Spectral Domain Optical Coherence Tomography |
| SLE | Slit Lamp Examination |
| TEAE | Treatment-Emergent AEs |
| TE SAE | Treatment-Emergent SAE |

Lineage Cell Therapeutics, Inc.
OpRegen® Protocol: CCN\_CT02 (Amendment #14)
Statistical Analysis Plan Version 1.0

12 October 2022

#### 2.0 INTRODUCTION

#### **General Overview**

CCN\_CT02 is a Phase I/IIa, multicenter, multinational open-label, interventional clinical trial of OpRegen®, a cell-based product composed of retinal pigment epithelium (RPE) cells, derived from human embryonic stem cells (hESCs) through a process of directed differentiation, which are implanted as a single administration to the worst vision eye of patients with advanced dry-form age-related macular degeneration (AMD) and geographic atrophy (GA) as a cell suspension (www.ClinicalTrials.gov Identifier: NCT02286089). The study involves dose escalation cohorts of targeted suspensions of 50x10³ to 200x10³ cells

methods of subretinal surgical administration of OpRegen were employed during the study; 1) pars planar vitrectomy (PPV) and retinotomy or, 2)

which utilized a sclerotomy and route to access the subretinal space.

#### Purpose of the Statistical Analysis Plan (SAP)

The purpose of this document is to provide a description of the statistical methods and procedures to be implemented for the analysis of data from the OpRegen clinical trial CCN-CT02. This document is based on protocol version amendment number 14, dated 9 April 2019. Any revisions to the SAP (both alternative and additional methods) will be made prior to database lock(s) and reasons for such revisions will be described in the final Clinical Study Reports (CSR).

#### 3.0 STUDY OBJECTIVES AND ENDPOINTS

## 3.1 Study Objectives

## 3.1.1 Primary Objectives

To evaluate the safety and tolerability of human embryonic stem cell-derived retinal pigment epithelium cells (OpRegen), transplanted subretinally to subjects with advanced dry age-related macular degeneration (AMD) with geographic atrophy (GA).

#### 3.1.2 Secondary Objectives

To evaluate the preliminary efficacy of OpRegen treatment by assessing the changes in ophthalmological parameters as measured by various methods of primary clinical relevance.



<sup>&</sup>lt;sup>1</sup> Refer to Section 2.3 in the <u>Investigator Brochure</u> for more information about the Product Description

## 3.2 Study Endpoints

## 3.2.1 Safety and Tolerability Endpoints

Safety and tolerability of OpRegen treatment will be assessed by:

- Incidence and frequency of treatment emergent adverse events (AEs)
- Treatment emergent changes in the following variable:
  - Ophthalmological evaluation:
    - ✓ Intraocular Pressure (IOP)



## 3.2.4 Efficacy Endpoints of Clinical Relevance

Preliminary efficacy assessments will utilize the below listed parameters:

- Directional change in the geographic atrophy (GA) lesion area over time
- Overall change in the GA lesion area of the study eye over time using SD-OCT and FAF
- Change from baseline over time in <u>BCVA</u> as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) chart
- Change from initial assessment over time in retinal sensitivity (as assessed by microperimetry)
- Change from baseline over time in Reading Speed Test
- Change from baseline over time in Low Luminance BCVA
- Correlation assessment between quantitative metrics derived from <u>FAF</u>, <u>SD-OCT</u> and <u>CFP</u> images
- Correlation assessment between functional and structural changes
- Change over time in National Eye Institute Visual Function Questionnaire-25 (<u>NEI VFQ-25</u>) Quality of Life (<u>QoL</u>) score
- Change over time in Functional Reading Independence (FRI) Index score

Statistical Analysis Plan Version 1.0

## 3.3 Study Hypothesis

As this is an open label, phase I/IIa dose escalation, safety, tolerability, and preliminary efficacy study, neither power assessment, nor formal hypotheses testing were planned for study outcome measures. However, for purposes of data analyses and this SAP, the Sponsor hypothesizes that implantation of OpRegen to subjects with advanced dry-form <u>AMD</u> with <u>GA</u> is safe, well-tolerated and provides evidence of preliminary efficacy based on pre-specified functional and structural assessments.

The primary hypothesis is that there will be no dose-limiting toxicity (<u>DLT</u>) and that implantation of OpRegen to subjects with progressive dry-form <u>AMD</u> with <u>GA</u> will be safe and well-tolerated. For this study <u>DLT</u> is defined as an <u>SAE</u> determined to be product related.

A secondary null hypothesis is that there will be no difference in disease progression, as measured by retinal function and structure, between the treated and untreated regions in the treated eye and between the treated and untreated eye of a subject.

#### 3.4 Study Assessments Schedules

Study assessments are described in detail in the protocol and summarized below in **Table 1**.

**Table 1. Study Assessments** 

| Assessment | Time points | Primary<br>Endpoints/<br>Safety | Efficacy Endpoints of<br>Clinical Relevance |
|---|---|---|---|
| Best-Corrected Visual Acuity (BCVA)-ETDRS Retro illuminated 4-meter ETDRS Chart "R" for refraction followed by Chart "1" and "2" BCVA is reported in number of letters read correctly. First, the right eye is tested with Chart 1 and then the left eye is tested with Chart 2. Must be conducted by trained examiner (technician acceptable) and as per "BCVA Instructions Manual". | # | V | 7 |
| Low Luminance Best Corrected Visual Acuity LL BCVA is measured by placing a 2.0-log-unit neutral density filter over the trial frame in front of the study eye and having the participant read the normally illuminated ETDRS chart using a different version of the chart. This test is optional as subjects with low vision will not be able to perform this test and is not applicable for Cohorts 1-3. | # | | <b>V</b> |
| Spectral Domain Optical Coherence Tomography (SDOCT) Images obtained by certified examiner (technician acceptable). Reading of images done by central reading center. Refer to Central Reading manual for instructions. | | V | V |
| | | V | |
| <b>Dilated Fundus Examination</b> (peripheral retina, macula, choroid, optic nerve, retinal/detachment, retinal or vitreous hemorrhage, vitreous hemorrhage density, vitreous cells.) | | V | |

| Assessment | Time points | Primary<br>Endpoints/<br>Safety | Efficacy Endpoints of<br>Clinical Relevance |
|---|---|---|---|
| Microperimetry Automated microperimetry to be performed in Cohort 3 (optional) and in Cohort 4. Must be conducted by certified examiner (technician is acceptable). Reading of images done by central reading center. Refer to Central Reading manual for instructions. | 4 | V | V |
| Fluorescein Angiography (FA) Standard procedure for detection of CNV. Must be conducted by certified examiner (technician is acceptable): at to verify dry AMD and absence of neovascular (wet) AMD, and on final exam at end of study; optional FA during follow-up in cases of suspected conversion to wet AMD | | V | |
| Intraocular Pressure (IOP) One IOP measurement per eye | • | V | |
| Slit Lamp Examination (Lids/Lashes, Conjunctiva, Cornea, Iris, Aqueous Cells, Aqueous Flare and Lens) Must be conducted by certified examiner (technician is acceptable) | | V | |
| Physical Examination including ECG, Vital Signs Clinical evaluation by the study-dedicated investigator or designee will be performed at several time points to evaluate pre- and post-implantation subject condition including immunosuppression treatment safety (see below)** | H | V | |
| Malignancy Assessment In the case of any suspected malignancies at screening, subject should be referred to appropriate medical specialist. | | √ | |
| Complete Blood count (including differential) / Chemistry (including Serum Electrolytes)/ Coagulation / Urinalysis | 4 | V | |
| Serology Assessment including testing for HIV, CMV, EBV, HBV and HCV | | √ | |
| | | V | |
| Immunology | | V | |

| Assessment | Time points | Primary<br>Endpoints/<br>Safety | Efficacy Endpoints of<br>Clinical Relevance |
|---|---|---|---|
| HLA-typing will be performed during or during one of the subsequent visits if not performed during | | | |
| | | V | |
| QuantiFERON (state of inoculation) To detect tuberculosis (TB) disease | | $\sqrt{}$ | |
| | 4 | V | |
| Fundus Autofluorescence Imaging (FAF) Images obtained by certified examiner (technician acceptable). Reading of images done by central reading center. Images are done by using blue light Heidelberg instrumentation. Each assessment for each subject must be done with the same camera used at Screening. Refer to Central Reading manual for instructions. | | V | <b>V</b> |
| Color Fundus Photography (CFP) Images obtained by certified examiner (technician acceptable). Reading of images done by central reading center. Color Images are done by using Zeiss instrumentation. Each assessment for each subject must be done with the same camera used at Screening. Refer to Central Reading manual for instructions. | | V | <b>V</b> |
| Reading Speed Test This test is mandatory for subjects are proficient in English. | | | V |
| NEI VFQ-25 Quality of Life (examiner version) 25 item subject reported outcome. Scores range from 0- 100 with the higher score indicating better visual function. | | | <b>V</b> |

| Assessment | Time points | Primary<br>Endpoints/<br>Safety | Efficacy Endpoints of<br>Clinical Relevance |
|---|---|---|---|
| Functional Reading Independence (FRI) Index The FRI index is a patient-reported outcome measure developed specifically for use in GA subjects. Scores derived from the index range from 1 (unable to do) to 4 (total independence) and may be analyzed as either categorical (which is preferred from a regulatory perspective) or continuous variables. This test should be administered in the subject's mother tongue language and is not applicable for Cohorts 1-3 | | | √<br> |

#### 4.0 STUDY DESIGN

Open-label, dose escalation study of 24 subjects with advanced dry-<u>AMD</u> and <u>GA</u> divided into four cohorts (<u>Figure 1</u>):

## Cohorts 1-3

The first 2 cohorts, consisted of 3 eyes of 3 legally blind subjects with best corrected visual acuity of 20/200 or less in the study eye, all received a single subretinal implantation of OpRegen.

The third cohort included 6 eyes of 6 subjects with best corrected visual acuity of 20/200 or less in the study eye, all received a single subretinal implantation of OpRegen.

Staggered intervals and safety data review by the independent data safety monitoring board (DSMB) occurred within and between cohorts to ensure subjects safety and welfare.

#### Cohort 4

The fourth cohort included 12 eyes from 12 subjects with <u>BCVA</u> between 20/64 and 20/250 in the study eye, all received a single subretinal targeted implantation of OpRegen.



Staggered intervals and safety data review by the <u>DSMB</u> occurred between at least the first two subjects of each delivery modality to ensure subject safety and welfare.



#### All Cohorts

The study is being conducted in participants with confirmed bilateral <u>GA</u> (Study Eye and Non-Study, Fellow Eye).

Figure 1. Protocol Enrollment Schema



#### 4.1 Definitions

#### 4.1.1 Study Day and Study Reference Period

Time will be measured as Study Day defined according to Clinical Data Interchange Standards Consortium (CDISC) standard. That is, the date of the OpRegen injection is study day can be calculated as follows:

Study Day = visit date – date of OpRegen injection

Last study day for a subject is the subject's last clinical visit date recorded on the subject status e<u>CRF</u>. If this date is missing for a subject, the last date found in the clinical database (e.g., clinical lab test date or date of vital sign collection) will be used as the last study date for the subject.

Total days on study are the total number of days a subject has been followed up after OpRegen injection. Mathematically it can be calculated as follows:

Total days on study = last study date – date of OpRegen injection + 1

#### 4.1.2 Baseline and Change from Baseline

Unless indicated otherwise, change from baseline (CFB) will be calculated as follows, where the baseline assessment is the last assessment before OpRegen injection:

CFB = Value at Visit - Baseline

Percent change from baseline (PCFB) will be calculated as follow:

PCFB (%) = 100\*(Value at Visit - Baseline)/Baseline

## 5.0 STUDY POPULATION

Subject characteristics, numbers, and all inclusion and exclusion criteria are described in Protocol Section 8.

#### 6.0 STATISTICAL ANALYSIS GENERAL CONSIDERATIONS

The planned sample size of 24 treated eyes, with targeted doses of  $50x10^3$  and up to  $200x10^3$  cells, is considered clinically appropriate for further characterization of the safety, tolerability, and preliminary efficacy of OpRegen in the treatment of subjects with advanced dry-form  $\underline{AMD}$  with  $\underline{GA}$ .

Comprehensive interim reports of accumulated safety, tolerability and preliminary available efficacy data were presented to the <u>DSMB</u> prior to escalation to the next to come study dose and to enrolment of the next to come study cohort. Between cohorts, and subjects when applicable, the next step to proceed occurred per <u>DSMB</u> recommendation based on accumulated safety data.

All measured variables and derived parameters will be listed individually and if appropriate, presented in summary tables by dose regimen group and overall, providing sample size, absolute and relative frequency for categorical variables, or sample size, arithmetic mean, standard deviation, median, minimum, and maximum for continuous variables. <u>Confidence interval</u>s will be presented for the efficacy endpoints for exploratory purposes only. Complete analyses to be prospectively performed are outlined in this SAP.

## 6.1 Analysis Sets

#### **All Treated Population**

The All Treated Population will include all subjects who received OpRegen. This will be used for all safety and efficacy analyses.

#### Per Protocol (PP) Analysis Set

The Per Protocol (PP) analysis set is a subset of the All Treated Analysis Set and will consist of all subjects who received the OpRegen implantation and violated none of the major protocol guidelines.

Statistical Analysis Plan Version 1.0

12 October 2022

## **6.2 Significance Level**

Though no formal hypothesis testing was originally planned for this study, for purposes of this SAP, a significance level of 0.05 using two-tailed tests will be utilized for any exploratory significance testing performed.

#### 6.3 Procedures for Handling Missing Data and Outliers

Missing or incomplete dates will be imputed per <u>Section 4.1.1</u> for the purposes of determining treatment emergence. All other missing data will not be imputed, unless otherwise noted.

All unscheduled visit data will be included in data listings. In the data summary tables, the presence of missing data will be indicated by the inclusion of a 'missing' category with categorical data, and a count and percentage of missing observations for continuous numeric data, where applicable.

## **6.4 Descriptive Statistics**

All measured variables and derived parameters will be listed individually and if appropriate, presented in summary tables by dose regimen group and overall, providing sample size, absolute and relative frequency for categorical variables, or sample size, arithmetic mean, standard deviation, median, minimum, and maximum for continuous variables. <u>Confidence interval</u>s will be presented for the efficacy endpoints for exploratory purposes only.

#### 7.0 STATISTICAL METHODS

All data collected for this study will be presented in summary tables, listings, and figures (TLFs) as indicated in <u>Section 11</u> of this SAP. Shells for TLFs with enough detail for programming will be provided as a guide to develop the programming SAS codes. These shells will be in sufficient detail to simulate the actual TLFs when they are created from the locked database.

Tabulations for continuous data will use a standard set of summary statistics: number of observations available (n), mean, standard deviation (SD), median, and range (minimum, maximum).

Categorical or dichotomous data will be tabulated using counts and percentages. The numerator and denominator for each percentage calculation will be specified in the footnotes of table shells.

Data listings will present all information recorded in e<u>CRF</u>s and any derived variable(s) included in the analysis datasets for all subjects and visits.

For the SAP primary hypothesis, the dose will be defined to exceed the maximally tolerated dose (MTD) if at least two of the subjects in a cohort have DLT.

If the dose has not exceeded the MTD in Cohort 1, the study will proceed to Cohort 2, pending the DSMB review. If the dose has not exceeded the MTD in Cohort 2, the study will proceed to Cohort 3, pending the DSMB review of data from Cohorts 1 and 2. Enrollment of Cohort 4, using either method of surgical delivery, will proceed only after review of the accumulated safety data by the DSMB.

For the SAP secondary hypothesis concerning changes in retinal structure and function following OpRegen implantation, the small number of subjects (3 per cohort in Cohorts 1 and 2, up to 6 in

Cohort 3 and approximately 12 in Cohort 4) precludes any definitive assessment of change through formal statistical testing. However, the following data analytical techniques will be used to describe the retinal structure and function results: assessing the changes in treated eyes will involve comparing the magnitude of observed changes in retinal structure and function to the distribution of changes between visits in a given subject (including historical data, when available), and will be also compared to the same measures gathered from previously studied populations of similarly affected subjects.

Measurements of retinal structure and function made on the non-treated eye of each subject will also be examined in the same way as for the treated eye to evaluate the extent to which placebo effects or unexpected temporal trends may be contributing to observed changes in retinal function.

## 7.1 Study Subjects

## 7.1.1 Subject Disposition

Subject disposition will be presented for the Screened Population. The following will be presented in a disposition table:

- Number of subjects screened
- Number of subjects dosed with OpRegen by cohort and overall (All Treated Population)
- Number and percentage of subjects who terminated prematurely before 1 Year Visit by cohort and overall
- Reason for premature termination before 1 Year Visit by cohort and overall
- Number and percentage of subjects who completed 1 Year Visit by cohort and overall

The number of subjects in the above categories will also be presented in a flow diagram figure.

A table with the number of screen failures and reason for screen failure will be produced.

#### 7.1.2 Protocol Deviations

A protocol deviation is any change, divergence, or departure from the study design or procedure defined in the protocol.

The following categories will be used to group protocol deviations:

- 1. Eligibility not met
- 2. Study Assessment Noncompliance
- 3. Other

The following are categorical reasons used to document why a protocol deviation occurred:

- 1. Subject illness
- 2. Clinical error
- 3. Investigator/staff decision
- 4. Other

Lineage Cell Therapeutics, Inc.

OpRegen® Protocol: CCN CT02 (Amendment #14)

Statistical Analysis Plan Version 1.0

12 October 2022

A subset of the protocol deviations can be identified as an important protocol deviation as described below:

Important Protocol Deviation: An important protocol deviation that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a subject's rights, safety, or well-being.

All documented protocol deviations in the study will be reviewed to identify all important protocol deviations by a data review team including representatives from clinical operations, medical, data management, and statistics.

A summary table of protocol deviations will be presented for the number and percentage of subjects in the following categories by cohort and overall:

- $\geq 1$  protocol deviation
- ≥1 important protocol deviation
- Important protocol deviation category
- Important protocol deviation reason
- Protocol deviation category
- Protocol deviation reason

#### 7.1.3 Demographics

A demographic and baseline characteristics table will be presented for the All Treated Population by cohort. The summary will include descriptive statistics for age, sex, race, weight, height, and BMI at baseline.

#### 7.1.4 Medical and Surgical History

At the ecretain and surgical procedures history will be recorded on the eCRF. Medical/Surgical History data will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) version 25.0 System Organ Class (SOC) and Preferred Term (PT).

#### 7.1.5 Concomitant Medications

All prior and concomitant medications, interventions and procedures will be tabulated. Prior and concomitant medications will be coded to the therapeutic drug classes and generic drug names using the World Health Organization Drug (WHODrug) classifications.

#### 7.1.6 Adverse Events

The collection period for adverse events for the purposes of this protocol begins once the subject has signed the informed consent form and ends after the will be listed by subject. The MedDRA (Version 25.0) will be used to classify all adverse events by SOC and PT.

A treatment emergent adverse event (<u>TEAE</u>) will be considered as any <u>AE</u> that starts on or after the date and time of the OpRegen administration, or if an <u>AE</u> that started before the OpRegen injection worsened after the administration of the investigational product.

A topline summary of treatment emergent adverse events with the number of events, number of subjects, and percentage of subjects for each category below will be tabulated by cohort.

- Any <u>TEAE</u> and <u>SAE</u>
- Subjects reporting at least one <u>TEAE</u> or <u>TE SAE</u> that is also related to OpRegen
- <u>TEAE</u> and <u>SAE</u> Severity: Grade 1/Mild, Grade 2/Moderate, Grade 3/Severe, Grade 4/Life Threatening/Disabling, Grade 5/Fatal
- Categories for all <u>TEAE</u> and with possible relationship to OpRegen

The following tables will be presented for the number of events by cohort:

- TEAE by preferred term sorted by descending number of overall events
- TEAE by SOC, PT\*
- TEAE by maximum severity\*
- TEAE by Possible Relationship to OpRegen\*

#### 7.1.7 Clinical Laboratory Tests

Summary statistics (N, mean, standard deviation, median, minimum, and maximum) will be tabulated for hematology, serum chemistry and urinalysis. For the minimum and maximum summary statistics, the minimum and maximum results taken during any assessment within cohort will be used.

#### 7.1.8 Vital Signs

Summary statistics (N, mean, standard deviation, median, minimum, and maximum) will be tabulated for vital sign parameters by cohort and overall. N will be calculated as the number of subjects with ≥1 assessment for the given parameter. For the minimum and maximum summary statistics, the minimum and maximum results taken during any assessment within cohort and overall will be used.

#### 7.1.9 Physical Exam

The number and percentage of subjects with abnormal physical exam results by system organ class at the will be tabulated by parameter for each cohort and overall.

## 7.1.10 Efficacy Analyses

All efficacy data will be listed for all subjects. Efficacy summaries will be presented for the Intent to Treat Population for all variables.

- Directional change in the geographic atrophy (GA) lesion area over time
- Overall change in the GA lesion area of the study eye over time using FAF
- Change from baseline over time in <u>BCVA</u> as measured by Early Treatment Diabetic Retinopathy Study (<u>ETDRS</u>) chart
- Change from baseline over time in Low Luminance <u>BCVA</u>
- Change from baseline over time in **IOP**

#### 8.0 GENERAL CONSIDERATIONS

In general, numerical variables in demographic and baseline characteristics will be summarized by displaying: n (non-missing sample size), mean, standard deviation, median, quartiles, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed

<sup>\*</sup>Subjects with >1 <u>AE</u> in respective category will only be counted once. For maximum severity tabulations, subjects will be counted once in the SOC and PT in the maximum severity.

levels will be reported for all categorical measures. Percentages will be calculated out of the total number of subjects per group.

Numerical effectiveness variables described above will be summarized displaying n, mean, median, standard deviation (SD), standard error (SE), quartiles, minimum, maximum.

All summary tables will be structured with a column for either treated or fellow eye.

No inferential statistics will be applied to baseline characteristics and safety variables unless specified otherwise.

In general, all data will be listed and sorted by treatment or fellow eye status, cohort number, site and subject, and when appropriate by visit number (or assessment date) as appropriate.

Most data manipulation, tables, figures, listings, and analysis will be documented in SAS programs and performed using  $SAS^{\mathbb{R}}$  Software version 9.4.

## 9.0 SEQUENCE OF PLANNED ANALYSES

Final analysis of safety and efficacy at the primary short-term endpoint (following last subject dosed)



An interim analysis will be performed using data from all subjects with a



Long-term follow-up analysis of safety and efficacy (5 years post-last OpRegen dose)

Final analysis will be performed using data from all subjects with a Year 5 post-treatment assessment.

#### 10.0 REPORTING CONVENTIONS

## **General reporting conventions**

All tables, listing and figures (TLFs) will be presented in portrait orientation, unless landscape orientation suggests that the information is easier to view. Legends will be used for all figures with more than one variable or item displayed. Figure lines should be wide enough to see the line after being copied.

All TLFs will have the name of the relevant SAS program (output name), the author, and a date-time stamp on the bottom of each output. All outputs will be produced on PDF to avoid changes during medical writing processes.

Titles should contain the following information:

- Output number
- Description of the data that is being summarized
- Type of analysis performed, and covariates used (if applicable)
- Analysis population

#### **Statistical summary conventions**

For tables, sample sizes for each treatment group will be presented as totals in the column header (N=x), where appropriate. Sample sizes shown with summary statistics are the number (n) of subjects with non-missing values.

Summaries for categorical variables will include only categories that subjects had a response in. Percentages corresponding to null categories (cells) will be suppressed. All summaries for continuous variables will include: N, mean, and <u>SD</u>. Other summaries (e.g. median, quartiles, 5%, 95% intervals, CV or %CV) will be used as appropriate. All percentages should be rounded and reported to a single decimal place (xx.x%). If percentages are reported as integers, percentages greater than 0% but <1% will be reported as <1%, whereas percentages greater than 99% but <100% will be reported as >99%. A percentage of 100% will be reported as 100%. No value of 0% should be reported. Any computation of percent that results in 0% is to be reported as a blank. P-values will be reported with three decimal places with a leading zero (0.001). P-values <0.001 will be reported as <0.001.

# 11.0 SUMMARY TABLES, FIGURES AND DATA LISTINGS

## **List of Tables**

| Table Number | Table Title |
|---|---|
| 14.1.1 | Subjects Disposition |
| 14.1.2 | Time in Study |
| 14.1.3 | Early Discontinuations |
| 14.1.4.1 | Demography screened subjects |
| 14.1.4.2 | Demography |
| 14.1.6 | Physical Examination |
| 14.1.7 | General Medical History |
| 14.1.8 | Concomitant Medications |
| 14.1.9 | Per Protocol Medications |
| 14.1.10 | AMD History |
| 14.1.11 | Ocular History |
| 14.1.5 | OpRegen Surgical Procedure |
| 14.3.1.1.1 | Frequency and Incidence of Treatment Emergent Adverse Events by MedDRA System Organ Class |
| 14.3.1.1.2 | Frequency and Incidence of Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term |
| 14.3.1.2.2 | Frequency and Incidence of Serious Treatment Emergent Adverse Events by MedDRA System Organ Class, Preferred Term |
| 14.3.1.4.2 | Frequency and Incidence of Treatment Emergent Adverse Events by Event Relationship to Per Protocol Treatment MedDRA System Organ Class, Preferred Term |
| 14.3.1.8.2 | Frequency and Incidence of Treatment Emergent Adverse Events by Ocular Toxicity MedDRA System Organ Class, Preferred Term |
| 14.3.1.9.2 | Frequency and Incidence of Treatment Emergent Adverse Events by Systemic Toxicity MedDRA System Organ Class, Preferred Term |
| 14.3.3.2 | Vital Signs |
| 14.3.2 | Laboratory results |
| 14.2.1 | Efficacy Geographic Atrophy |
| 14.2.2 | Efficacy Best Corrected Visual Acuity |
| 14.2.3.1 | Efficacy Intra-Ocular Pressure |

Lineage Cell Therapeutics, Inc.
OpRegen® Protocol: CCN\_CT02 (Amendment #14)
Statistical Analysis Plan Version 1.0

12 October 2022

# **Figures**

| Figure Number | Figure Title |
|-------------------|------------------------------------------------|
| Figure 14.1.1 | Subject Disposition Tree All Screened Subjects |
| Figure 14.3.3.1 | Vital signs |
| Figure 14.3.2.1-7 | Laboratory |
| Figure 14.2.1.1 | Efficacy Geographic Atrophy |
| Figure 14.2.1.2 | Efficacy Geographic Atrophy Annual rate |
| Figure 14.2.2 | Efficacy Best Corrected Visual Acuity |
| Figure 14.2.3 | Efficacy Intra-Ocular Pressure |

## **Data Listings**

| <b>Listing Number</b> | Listing Title |
|-----------------------|--------------------------------------------------|
| 16.1.1.1 | Subject Disposition |
| 16.1.2 | Subjects Time in Study |
| 16.1.3 | Early Discontinuations |
| 16.1.4 | Demography |
| 16.1.6 | Physical Examination |
| 16.1.7 | General Medical History |
| 16.1.8 | Concomitant Medications |
| 16.1.9 | Per Protocol Medications |
| 16.1.10 | AMD History |
| 16.1.11 | Ocular History |
| 16.1.5 | OpRegen Surgical Procedure |
| 16.3.1.1 | Treatment Emergent Adverse Events |
| 16.3.1.3 | Serious Adverse Events |
| 16.3.1.5 | Adverse events outcome classified as Fatal/Death |
| 16.3.3 | Vital signs |
| 16.3.2 | Laboratory Results |
| 16.2.1.1 | Efficacy Geographic Atrophy |
| 16.2.1.2 | Efficacy Geographic Atrophy Annual rate |
| 16.2.2 | Efficacy Best Corrected Visual Acuity |
| 16.2.3 | Efficacy Intra-Ocular Pressure |